CLINICAL TRIAL: NCT00822263
Title: The Use of Anti-oxidants to Reduce Sequela of Mild TBI (mTBI) After Blast Exposure
Brief Title: The Use of Anti-oxidants to Reduce Sequela of Mild Traumatic Brain Injury (mTBI) After Blast Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Michael E. Hoffer, CAPT MC USN, U.S. Military
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNC-IRAQ-08-040
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2009-01

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mild traumatic brain injury; anti-oxidant; early treatment
MeSH Terms: conditions — Brain Concussion | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): control
  Interventions: Drug: Placebo
- 1 (Experimental): Active medicine
  Interventions: Drug: N-acetyl-cysteine (NAC)

INTERVENTIONS:
Drug: N-acetyl-cysteine (NAC) — Anti-oxidant in a pill format
  Arms: 1
Drug: Placebo — Control for study
  Arms: 2

SUMMARY:
The administration of N-acetyl-cysteine (an anti-oxidant) for seven days along with observation will result in improved hearing and balance function in individuals who demonstrate these disorders after blast exposure when compared to a placebo medicine and observation at the seven day time point.

DETAILED DESCRIPTION:
5.0 RESEARCH PLAN: The goal of this study is to examine the use of one anti-oxidant, N acetylcysteine (NAC), in individuals who suffer blast injury and demonstrate early sequela of mTBI.

Recent changes in war fighting and operational situations have changed the injury patterns that our troops face in all aspects of military operations. Mild traumatic brain injury (mTBI) is among the most common injuries seen in the current theater of operations. While other injury patterns have shown a decrease over the last twelve months, mTBI from blast exposure has continued to be seen at increasing levels. This may be due in part to the fact that research has shown the individuals may suffer mTBI secondary to blast injury from one significant exposure or from repeated low level exposure which is more common as individuals rotate back to the theatre of operations for second, third, and even forth tours of duty. The sequela of mTBI include balance disorders, hearing loss, and cognitive dysfunction. These disorders can present immediately after the injury or several weeks after the injury but tests of function can detect injury shortly after the injury. Evidence exists in laboratory work and in human studies that anti-oxidant medicine can reduce/eliminate the sequela of mTBI if administered within 8-24 hours of injury.

5.1 OBJECTIVES: A population and single-subject design, double blinded, placebo controlled study comparing the effectiveness of the observation and administration of the anti-oxidant NAC to placebo in individuals suffering the sequela of mTBI after a single or multiple blast exposures.

5.2 HYPOTHESIS: The administration of NAC for seven days along with observation will result in improved hearing and balance function in individuals who demonstrate these disorders after blast exposure when compared to a placebo medicine and observation at the seven day time point

5.3 SPECIFIC AIMS:

1. To determine the frequency of hearing loss and balance disorders in those exposed to blast injury that have non-emergent or non-urgent medical or surgical disorders and display a pattern of injury consistent with mTBI.
2. To determine the effectiveness of one week of anti-oxidant, N-acetylcysteine combined with observation, in the reduction of hearing loss and balance disorders one week after injury as compared to placebo medication and observation.
3. To determine the effectiveness of one week of anti-oxidant, N-acetylcysteine combined with observation, in the reduction of hearing loss and balance disorders six months after injury as compared to one week of placebo medication and observation.

ELIGIBILITY:
Inclusion Criteria:

1. Be active duty United States Service member
2. Be between the ages of 18 and 50 years
3. Present to TQ Surgical within 24 hours of blast exposure.
4. Have complains consistent with possible TBI including hearing loss, dizziness, lightheadedness, cognitive difficulties, and/or had loss of consciousness.
5. Are not expressly excluded by the criteria listed below.

Exclusion Criteria:

1. Require urgent or emergent surgical procedures.
2. Will require medical evacuation to any level III or higher facility (other then to a level III for a CT scan only).
3. Has evidence of an open head wound.
4. Pregnant Females
5. The use, within the last seven days, of a nutritional supplement containing an anti-oxidant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Relief of symptoms of mTBI | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Hoffer, M.D., Principal Investigator — U.S. Military
Locations (1):
- TQ Surgical, AL Taqaddum, Iraq

REFERENCES:
- [Derived] Hoffer ME, Balaban C, Slade MD, Tsao JW, Hoffer B. Amelioration of acute sequelae of blast induced mild traumatic brain injury by N-acetyl cysteine: a double-blind, placebo controlled study. PLoS One. 2013;8(1):e54163. doi: 10.1371/journal.pone.0054163. Epub 2013 Jan 23. PMID 23372680